CLINICAL TRIAL: NCT06734520
Title: Clinical Study of Super Transplantation in the Treatment of Severe β-thalassemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024217A01
Record Dates: First submitted 2024-11-16; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Thalassemia Majors (Beta-Thalassemia Major); Haplo-identical Donors
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Severe β -thalassemia (Experimental): Children with β-thalassemia major received super transplantation, and chimerism tests were performed at 3 months, 6 months, 9 months, and 1 year after transplantation to evaluate the safety and effectiveness.
  Interventions: Drug: super-transplantation in 3 severe β -thalassemia pediatric patients.

INTERVENTIONS:
Drug: super-transplantation in 3 severe β -thalassemia pediatric patients. — Haplo-identical donors are mobilized with G-CSF and PBMCs that contain CD34+ stem cells and CD3+ lymphocytes will be extracted by blood cell separators. Then the patients will be infused with the PBMC

SUMMARY:
This is a single-arm, open label, phase 1 study in subjects with beta-thalassemia. This study will evaluate the safety and efficacy of preconditioning-free super-transplantation on beta-thalassemia pediatric patients.

DETAILED DESCRIPTION:
Patient screening:

1. Two months before transplantation, pediatric patients are evaluated by our center, and the patients meeting the inclusion criteria will be screened into the group.
2. Investigators and doctors will give detailed information about the benefits and risks of participating in the study, and the informed consents are further signed.

Transplant conduction:

1. Donor mobilization: HLA-fully matched or haplo-identical donors are mobilized subcutaneously for five days with human granulocyte colony-stimulating factor (G-CSF) and the peripheral blood mononuclear cells (PBMCs) that contain a certain numbers of CD34+ stem cells and CD3+ lymphocytes will be extracted by blood cell separators.
2. Transplant regimen: Hydroxycarbamide will be used to reduce the total white blood cells before transplant. However, no traditional transplantation conditioning will be performed, including but not limited to busulfan, fludarabine, Cyclophosphamide, ATG, and irradiation. Splenectomy should be performed if the longitudinal diameter of the spleen exceeds the normal value by 4 cm.
3. Cell infusion: Pediatric patients will be infused with the PBMCs intravenously at day 0.
4. GVHD prophylaxis: The dosage of immunosuppressants is half of the conventional post-transplantation level, but adjustments to the dosage may be necessary based on specific circumstances.
5. Infection management: Antibacterial, antifungal medications, and anti-Pneumocystis medications need to be administered during the period of granulocytopenia. The preemptive treatment for cytomegalovirus will be performed when the virus serological test is positive.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of severe β -thalassemia
2. Age between 7-10 years old, male and female; Weight < 40kg
3. The patient has or does not have an HLA-compatible or semi-compatible donor, but unconditional transplantation or refusal of blood stem cell transplantation; Patients with thalassemia gene therapy without conditions or refusal;
4. There are fully compatible or incompatible HLA donors, and the physical examination meets the donor conditions;
5. The patient and family members agree to receive hypertransplant therapy and sign a written informed consent prior to the transplant trial.

Exclusion Criteria:

1. Mental patients;
2. Participants in other drug clinical trials within the past 1 month;
3. There are no suitable HLA-incompatible donors.
4. Other researchers decide that it is not suitable to participate in this researcher.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
chimeric status | 1 year after transplantation.
  Detecting the chimerism in recipients' peripheral blood and bone marrow.Chimerism is generally measured in percentages(%)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, PHD, Study Director — Guangzhou Medical University Affiliated Women's and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center Affiliated to Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Share IPD with 5th Medical Center ofA General Hospital
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The start date is October 2024 and the end date is July 2029
Access Criteria: The sponsors and collaborators are able to access the IPD and supporting information, IPD relies on team collaboration , as well as continuous improvement in innovation and efficiency. Participants will share project information, including the project's objectives, statistical datas, and clinical study report.

REFERENCES:
- [Background] Ali S, Mumtaz S, Shakir HA, Khan M, Tahir HM, Mumtaz S, Mughal TA, Hassan A, Kazmi SAR, Sadia, Irfan M, Khan MA. Current status of beta-thalassemia and its treatment strategies. Mol Genet Genomic Med. 2021 Dec;9(12):e1788. doi: 10.1002/mgg3.1788. Epub 2021 Nov 5. PMID 34738740
- [Background] Shafique F, Ali S, Almansouri T, Van Eeden F, Shafi N, Khalid M, Khawaja S, Andleeb S, Hassan MU. Thalassemia, a human blood disorder. Braz J Biol. 2021 Sep 3;83:e246062. doi: 10.1590/1519-6984.246062. eCollection 2021. PMID 34495151
- [Background] Dever DP, Bak RO, Reinisch A, Camarena J, Washington G, Nicolas CE, Pavel-Dinu M, Saxena N, Wilkens AB, Mantri S, Uchida N, Hendel A, Narla A, Majeti R, Weinberg KI, Porteus MH. CRISPR/Cas9 beta-globin gene targeting in human haematopoietic stem cells. Nature. 2016 Nov 17;539(7629):384-389. doi: 10.1038/nature20134. Epub 2016 Nov 7. PMID 27820943